CLINICAL TRIAL: NCT04841733
Title: Evaluation of the Effectiveness of the Combination of Different Post-effort Recovery Methods on Quality and Recovery Time in Semi-professional Soccer Players
Brief Title: Effectiveness of Recovery Protocols Combination in Soccer Players
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Vic - Central University of Catalonia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: RCTREC002
Record Dates: First submitted 2021-04-08; First posted 2021-04-12 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Soccer; Physical Stress; Fatigue
Keywords: Performance; Recovery; Fatigue; Soccer
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Protocol I: Foam Roller (FR) + Cold-Water Immersion (CWI) (Experimental): Foam Roller (FR) Cold-Water Immersion (CWI)
  Interventions: Other: Foam Roller (FR); Other: Cold-Water Immersion (CWI)
- Protocol II: Stretching (STR) + Cold-Water Immersion (CWI) (Experimental): Stretching (STR) Cold-Water Immersion (CWI)
  Interventions: Other: Stretching (STR); Other: Cold-Water Immersion (CWI)
- Protocol III: Foam Roller (FR) + Stretching (STR) (Experimental): Foam Roller (FR) Stretching (STR)
  Interventions: Other: Foam Roller (FR); Other: Stretching (STR)
- Protocol IV: Foam Roller (FR) + Stretching (STR) + Cold-Water Immersion (CWI) (Experimental): Foam Roller (FR) Stretching (STR) Cold-Water Immersion (CWI)
  Interventions: Other: Foam Roller (FR); Other: Stretching (STR); Other: Cold-Water Immersion (CWI)

INTERVENTIONS:
Other: Foam Roller (FR) — Foam Roller (FR): participants will follow the Foam Roller protocol using a polyvinylchloride pipe roller (10.3-cm diameter, 0.3-cm thickness surrounded by a 1,5-cm thickness neoprene foam). They will begin with the Foam Roller at the most proximal portion of the muscle and to roll as much body mass as tolerable back and forth along it as smoothly as possible at a cadence of 1 second superior and 1 second inferior as determined with the metronome. Foam Roller will be performed for 45 seconds followed by a 15-second rest for each muscle group (quadriceps, adductors, hamstrings, abductors and calf) in each extremity and repeated once.
  Arms: Protocol I: Foam Roller (FR) + Cold-Water Immersion (CWI); Protocol III: Foam Roller (FR) + Stretching (STR); Protocol IV: Foam Roller (FR) + Stretching (STR) + Cold-Water Immersion (CWI)
Other: Stretching (STR) — Stretching (STR): participants will perform 8-min of static stretching, involving 3 bilateral repetitions of 30 seconds held stretches to the quadriceps, adductors, hamstrings, abductors and calf muscles.
  Arms: Protocol II: Stretching (STR) + Cold-Water Immersion (CWI); Protocol III: Foam Roller (FR) + Stretching (STR); Protocol IV: Foam Roller (FR) + Stretching (STR) + Cold-Water Immersion (CWI)
Other: Cold-Water Immersion (CWI) — Cold-Water Immersion (CWI): will be the last strategy used. Participants will immerse their lower body to the level of the hips for 10 minutes in cold water (10° C).
  Arms: Protocol I: Foam Roller (FR) + Cold-Water Immersion (CWI); Protocol II: Stretching (STR) + Cold-Water Immersion (CWI); Protocol IV: Foam Roller (FR) + Stretching (STR) + Cold-Water Immersion (CWI)

SUMMARY:
The main objective of this project is to compare the effectiveness of combining different recovery methods on perceptual and physical performance on soccer players.

DETAILED DESCRIPTION:
A crossover study will be performed and players will be assigned to different recovery methods combinations after their participation in a football game. The investigators will take baseline measures before the game and post-competition measures 24 hours after the game (one hour before the recovery intervention). Moreover, another two measure moments will be used, 24 and 48 hours after the recovery intervention.

ELIGIBILITY:
Inclusion Criteria:

* semi-professional soccer players
* 75 minutes game participation (minimum)
* 5 years of experience practicing soccer

Exclusion Criteria:

* goalkeepers
* injured players

Min Age: 16 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-04-18 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Neuromuscular or physical performance measures change: jump height | Baseline, 1 hour before intervention, 24 hours after intervention, 48 hours after intervention
  Counter Movement Jump (CMJ) will be performed to determine the maximum height in centimeters (cm). From standing position with the hands fixed on the hips, participants will be required to bend their knees to a freely chosen angle and perform a maximal vertical jump. Participants will be instructed to keep their body vertical throughout the jump, and to land with knees fully extended. Any jump that will be perceived to deviate from the required instructions will be repeated. Players will jump 3 times as high as possible and the best attempt will be used in subsequent analysis. A 15-s passive recovery phase will be provided between jumps.
Neuromuscular or physical performance measures change: jump flight and contact time | Baseline, 1 hour before intervention, 24 hours after intervention, 48 hours after intervention
  Counter Movement Jump (CMJ) will be performed to determine the jump flight and contact time in milliseconds (ms). From standing position with the hands fixed on the hips, participants will be required to bend their knees to a freely chosen angle and perform a maximal vertical jump. Participants will be instructed to keep their body vertical throughout the jump, and to land with knees fully extended. Any jump that will be perceived to deviate from the required instructions will be repeated. Players will jump 3 times as high as possible and the best attempt will be used in subsequent analysis. A 15-s passive recovery phase will be provided between jumps.

SECONDARY OUTCOMES:
Subjective perceptual/well-being questionnaire measures change | Baseline, 1 hour before intervention, 24 hours after intervention, 48 hours after intervention
  The well-being questionnaire (McLean et al. 2010) will assess participants' fatigue, sleep quality, general muscle soreness, stress levels and mood on a five-point scale (scores of 1[worst outcome] to 5 [best outcome], 0.5 point increments). Overall well-being will then be determined by summing the five scores.
Total Quality Recovery perceived (TQRper) scale. Subjective perceptual questionnaire measures change | Baseline, 1 hour before intervention, 24 hours after intervention, 48 hours after intervention
  Players will be asked to rate their recovery using the subjective questionnaire Total Quality Recovery perceived (TQRper) scale (Kenttä & Hassmén, 1998) answering the question "how recovered you feel?" on a scale which ranges from 0 (very poorly recovered) to 10 (very well recovered) and it's used as a subjective measurement to assess the fatigue suffered by the players (Laurent et al., 2011).
Rate of Perceived Exertion (RPE) scale. Subjective perceptual questionnaire measures change | Baseline, 1 hour before intervention, 24 hours after intervention, 48 hours after intervention
  Players will be asked to rate their rate of perceived exertion using Rate of Perceived Exertion (RPE) Borg's scale answering the question "how exhausted do you feel?" on a scale which ranges from 0 (extremely well-rested) to 10 (extremely exhausted) (Casamichana et al., 2013).

CONTACTS AND LOCATIONS:
Overall Officials: Albert Altarriba-Bartes, Principal Investigator — UVic-UCC
Locations (1):
- Universitat de Vic-Universitat Central de Catalunya, Vic, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McLean BD, Coutts AJ, Kelly V, McGuigan MR, Cormack SJ. Neuromuscular, endocrine, and perceptual fatigue responses during different length between-match microcycles in professional rugby league players. Int J Sports Physiol Perform. 2010 Sep;5(3):367-83. doi: 10.1123/ijspp.5.3.367. PMID 20861526
- [Background] Kentta G, Hassmen P. Overtraining and recovery. A conceptual model. Sports Med. 1998 Jul;26(1):1-16. doi: 10.2165/00007256-199826010-00001. PMID 9739537
- [Background] Laurent CM, Green JM, Bishop PA, Sjokvist J, Schumacker RE, Richardson MT, Curtner-Smith M. A practical approach to monitoring recovery: development of a perceived recovery status scale. J Strength Cond Res. 2011 Mar;25(3):620-8. doi: 10.1519/JSC.0b013e3181c69ec6. PMID 20581704
- [Background] Casamichana D, Castellano J, Calleja-Gonzalez J, San Roman J, Castagna C. Relationship between indicators of training load in soccer players. J Strength Cond Res. 2013 Feb;27(2):369-74. doi: 10.1519/JSC.0b013e3182548af1. PMID 22465992